CLINICAL TRIAL: NCT05794256
Title: A Prospective Analysis of the Gender Specific Role of Steroid Hormones on the Outcome on Patients After Polytrauma
Brief Title: Genderspecific Differences in Hormone Levels After Trauma
Acronym: SteroPoly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-687-S-SR
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2022-11

CONDITIONS: Polytrauma
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions are planned — No interventions are planned

SUMMARY:
The goal of this prospective study with the aim to establish a registry is to learn about the role of steroid hormones in severely injured patients. The main question it aims to answer is whether steroid hormones influence morbidity and mortality after severe trauma.

This is a prospective study with the aim to establish a large registry for severely injured patients and their hormonal status.

Hormone levels will be measured upon arrival in the emergency room and within the following few days after trauma. Furthermore a detailed questionnaire aims to answer any hormone-related health questions.

ELIGIBILITY:
Inclusion Criteria:

* Polytrauma with ISS≥16,
* severe traumatic brain injury (AIS ≥3)
* over the age of 18
* must reach emergency room alive

Exclusion Criteria:

* pregnant patients
* dead on arrival to the hospital
* incarcerated patients
* secondarily transferred patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients suffering from severe trauma (ISS ≥ 16) or severe traumatic brain injury (AIS ≥3) will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-18 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | within 1 year after trauma

CONTACTS AND LOCATIONS:
Locations (1):
- Technical University Munich, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No